CLINICAL TRIAL: NCT03559907
Title: Partnering for Prevention: Building Healthy Habits in Underserved Communities
Acronym: P4P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Principal Investigator, Angela Caldwell, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO17080038
Record Dates: First submitted 2018-05-15; First posted 2018-06-18 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Parenting; Child Nutrition Disorders
Keywords: prevention; nutrition; early childhood; parent training; underserved
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Quasi-Experimental: Three community sites will be randomized to receive on of three prevention interventions:
  1. Cooking Matters for Parents
  2. Promoting Routines of Exploration and Play during Mealtime (Mealtime PREP)
  3. Combined (Cooking Matters + Mealtime PREP)
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors who are rating intervention fidelity will be blinded to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cooking Matters for Parents (Experimental): Trained instructors with a background in nutrition or culinary arts will lead six weekly, two-hour sessions to groups of 10 parent participants at local Family Support Centers.
  Interventions: Behavioral: Cooking Matters for Parents
- Mealtime PREP (Experimental): Trained group leaders with experience in pediatric occupational therapy will lead six weekly, two-hour, Mealtime PREP sessions to groups of 10 parent participants at local Family Support Centers.
  Interventions: Behavioral: Mealtime PREP
- Cooking Matters + Mealtime PREP (Experimental): Parents will receive both programs in succession. They will attend Cooking Matters for Parents followed by Mealtime PREP. In total, this will equal 12 weekly, two-hour sessions delivered to groups of 10 parent participants at a local Family Support Center.
  Interventions: Behavioral: Cooking Matters for Parents; Behavioral: Mealtime PREP

INTERVENTIONS:
Behavioral: Cooking Matters for Parents — Cooking Matters for Parents focuses on teaching parents of young children important lessons about self-sufficiency in the kitchen. Participants have the opportunity to practice fundamental lessons including knife skills, reading ingredient labels, cutting up a whole chicken, and making a healthy meal for a family of four on a budget of ten dollars. Each session includes meal preparation, didactic teaching, and sharing the meal as a group. Instructors share their education and experience and discuss how to choose healthy, affordable fruits and vegetables at the grocery store. Each week, adults take home a bag of groceries after each class so they can practice the recipes taught that day.
  Arms: Cooking Matters + Mealtime PREP; Cooking Matters for Parents
Behavioral: Mealtime PREP — Parents are trained to deliver each intervention component during mealtimes using a step-wise, behavioral activation approach. The parent-training prong of the Mealtime PREP intervention incorporates four active ingredients of behavioral activation (1. skills training; 2. goal-setting; 3. activity scheduling; and 4. activity monitoring) to help parents build a family meal routine that is enriched with techniques to promote child food acceptance. Each week, parents will take home healthy groceries to practice making healthy snacks and side dishes in the home.
  Other Names: Promoting Routines for Exploration and Play during Mealtime
  Arms: Cooking Matters + Mealtime PREP; Mealtime PREP

SUMMARY:
This pilot study will estimate the unique and additive benefits of two parent-training programs (Cooking Matters for Parents and Promoting Routines of Exploration and Play during Mealtime) offered in undeserved communities.

DETAILED DESCRIPTION:
The overall purpose of this research study is to estimate the nutritional benefits (in terms of intake and variety) of the Mealtime PREP intervention, as compared to, and in combination with nutrition education programming being offered in underserved neighborhoods of the greater Pittsburgh area. This project will examine the effects of Mealtime PREP groups as compared with established nutrition education groups, Cooking Matters for Parents. More importantly, this study will determine if offering these interventions in combination offers greater benefits than each in isolation. There are two specific aims of this pilot trial.

1. To examine the effects of a combined program (Cooking Matters + Mealtime PREP) in comparison to offering each of these programs (Cooking Matters vs. Mealtime PREP) in isolation on child nutrition over time.
2. To explore the effects of each of these programs (Cooking Matters vs. Mealtime PREP) and the combined program (Cooking Matters + Mealtime PREP) on parental stress and parent/child interaction over time.

The investigators predict that children in all three arms (Cooking Matters, Mealtime PREP, and Cooking Matters + Mealtime PREP) will demonstrate improved nutrition. The investigators also predict that participants who receive the Mealtime PREP intervention will demonstrate better stability of gains over time.

ELIGIBILITY:
Inclusion Criteria:

* Parent to a child aged 1-5 years
* Speaks English
* Willing to participate in 6 or 12 weekly group sessions at local Family Support Center

Exclusion Criteria:

* Previously completed a Cooking Matters for Parents cooking class

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline 3-Day Food Diary (dietary variety) at 6 months | 6 months
  The 3-Day Food Diary is the preferred method of dietary assessment (intake and variety of food consumed) because of a balance between validity and burden. Includes all food consumed and approximate servings for 3 days.Frequencies of foods consumed from different food groups and basic nutritional intake related to the numbers of servings of food in each food group consumed will be calculated. Servings in each category will be compared to national daily recommendations.

SECONDARY OUTCOMES:
Change from Baseline Nutrition Screening Tool for Every Preschooler (nutritional risk) at 6 months | 6 months
  17 item, validated screen for young children (1-5 years) that categorizes risk of nutritional problems into 3 categories (score range = 1 (minimum) - 68 (maximum); 1 - 20 = low risk, 21-25 = moderate risk, and 26+ = high risk). Higher scores indicate higher risk for nutritional problems (i.e. lower scores are better).
Change from Baseline Parenting-Stress Inventory, Short-Form (PSI-SF) at 6 months | 6 months
  36 item scale validated in a sample of low-income families with preschoolers to assess parental stress in three domains and overall. Raw scores are converted to percentiles for interpretation using this tool. For the total parenting stress score, and all three domain scores (Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child), higher percentiles are interpreted as higher stress (range =1-99%) with scores >90% indicating clinically significant levels of parenting stress.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Caldwell, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caldwell AR, Terhorst L, Krall JS, Thum DW, Uman HR, Dodd JL, Haus EE, Bendixen RM. Partnering for prevention in under-resourced communities: a randomized pilot study. Nutr J. 2022 Nov 25;21(1):72. doi: 10.1186/s12937-022-00824-7. PMID 36434698